CLINICAL TRIAL: NCT06777563
Title: Ecological Momentary Assessment Combined mHealth-based Psychosocial Intervention to Prevent Postpartum Depression in Pregnant Women: a Pilot Randomized Controlled Trial
Brief Title: EMA and mHealth in Preventing Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PPD prevention
Record Dates: First submitted 2025-01-07; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Postpartum Depression (PPD); Ecological Momentary Assessment; mHealth Intervention
Keywords: postpartum depression; ecological momentary assessment; mHealth-based intervention; pregnant women
MeSH Terms: conditions — Depression, Postpartum | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (EMA + IM) (Experimental): The EMA+IM group (group A) will receive an evidence-based intervention composed of brief psychological counselling and health education, 2-week EMA, 10-week mHealth-based psychological support, and CBT-guided telephone counselling, guided by comprehensive assessment.
  Interventions: Behavioral: Brief psychological counselling and health education; Behavioral: 2 Weeks of Ecological Momentary Assessment (EMA); Behavioral: 10 weeks of mobile health psychological support; Behavioral: CBT-guided telephone counselling booster
- EMA group (Experimental): The EMA group (Group B) will receive brief psychological counselling and health education and 2-week EMA.
  Interventions: Behavioral: Brief psychological counselling and health education; Behavioral: 2 Weeks of Ecological Momentary Assessment (EMA)
- Control group (Active Comparator): The control group (group C) will receive only brief psychological counselling and health education.
  Interventions: Behavioral: Brief psychological counselling and health education

INTERVENTIONS:
Behavioral: Brief psychological counselling and health education — This is a brief 1-on-1 psychological counselling, including potential mood fluctuation during pregnancy, possible prepartum depressive symptoms, and available psychiatric consultation and medication in Hong Kong with self-help psychoeducational materials.
Behavioral: 2 Weeks of Ecological Momentary Assessment (EMA) — The 2-week EMA period will start the next day. Participants will be prompted to answer questions about emotion (e.g. worry, enjoyment, anxiety, etc.) and other lifestyle and environmental triggers through the smartphone notification function. There will be a 2-hour window for each assessment before expiration and total 5 assessments a day.
  Arms: EMA group; Intervention group (EMA + IM)
Behavioral: 10 weeks of mobile health psychological support — A total of 20 regular instant messages (e.g., via WhatsApp) personalised by baseline demographic characteristics (current pregnancy details, history of postpartum mental illness) and results of EMA will be sent to the participants in multi-media formats.
  Arms: Intervention group (EMA + IM)
Behavioral: CBT-guided telephone counselling booster — A 45-minute telephone counselling based on CBT.
  Arms: Intervention group (EMA + IM)

SUMMARY:
This proposed study aims to develop and examine the feasibility, acceptability, and preliminary effectiveness of a proactive intervention model that combines brief psychological counselling, Ecological Momentary Assessment (EMA), mHealth-based psychological support, and CBT-guided telephone counselling to prevent postpartum depression (PPD).

DETAILED DESCRIPTION:
The target participants are pregnant women between 20 and 28 weeks of gestation with a total EPDS-10 score of ≥7. Sixty participants will be actively recruited from the Department of Obstetrics and Gynaecology at Queen Mary Hospital (QMH), a major acute hospital in Hong Kong. Recruitment will extend to other public hospitals if needed.

This study will be a three-arm (allocation ratio:1:1:1; permutated block size of 3, 6, and 9), single-blinded, parallel, pilot randomised controlled trial (RCT) with follow-ups at 2, 4, 6, and 8 weeks post-enrollment using standard methodology (CONSORT) to evaluate the effectiveness of the intervention. The EMA+IM group (group A) will receive an evidence-based intervention composed of brief psychological counselling and health education, 2-week EMA, mHealth-based psychological support, and CBT-guided telephone counselling, guided by comprehensive assessment. The EMA group (Group B) will only receive a 2-week EMA, and the control group (group C) will receive only brief psychological counselling and health education. Surveys will be collected via telephone after childbirth. Semi-structured individual interviews will be conducted with the participants in the intervention group to understand the experience and the perceptions towards the EMA data collection and mHealth-based intervention on mental health.

The primary clinical outcome of this study will be the difference in the EPDS scores between the two groups at 2 weeks postpartum. Secondary clinical outcomes will include differences in anxiety levels, stress levels, and insomnia symptoms at 2, 4, 6 and 8 weeks postpartum. Differences in participants' self-rated health, family functioning, family well-being and perceived happiness will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women who are in their 20 to 28 weeks of gestation,
2. Receiving regular antenatal care service in Hong Kong,
3. Had a total score ≥7 in EPDS-10 (suggesting potential distress symptoms),
4. Able to read and understand Chinese and use an instant messaging app weekly

Exclusion Criteria:

1) Pregnant women who are undergoing psychiatric/psychological treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Postpartum depression | 2-week postpartum
  Postpartum depression will be measured by Edinburgh Postnatal Depression Scale (EPDS-10). The score ranges from 0-30. 0-9 indicates minimal or no depressive symptoms.10-12 suggests mild depressive symptoms and further monitoring may be recommended.13-14 indicates moderate depressive symptoms and a potential need for further assessment.15-30 suggests significant depressive symptoms and likely clinical depression, requiring further evaluation and intervention.

SECONDARY OUTCOMES:
Postpartum depression | 4, 6, 8 weeks postpartum
  Postpartum depression will be measured by the Edinburgh Postnatal Depression Scale (EPDS-10). The score ranges from 0-30. 0-9 indicates minimal or no depressive symptoms.10-12 suggests mild depressive symptoms and further monitoring may be recommended.13-14 indicates moderate depressive symptoms and a potential need for further assessment.15-30 suggests significant depressive symptoms and likely clinical depression, requiring further evaluation and intervention.
Anxiety | 2, 4, 6, 8 weeks postpartum
  Anxiety will be measured by the 7-item Generalized Anxiety Disorder (GAD-7). The total score ranges from 0 to 21. A higher score on the GAD-7 indicates greater severity of anxiety symptoms.
Depression | 2, 4, 6, 8 weeks postpartum
  Depression will be measured by the 9-item Patient Health Questionnaire (PHQ-9). The total score ranges from 0 to 27. A higher score on the PHQ-9 indicates greater severity of depressive symptoms.
Stress | 2, 4, 6, 8 weeks postpartum
  Self-perceived stress will be measured by the 10-item Perceived Stress Scale (PSS-10). The total score ranges from 0 to 40. A higher score on the PSS-10 indicates greater perceived stress, reflecting a higher level of distress or difficulty in managing life's challenges.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - School of Nursing, The University of Hong Kong, Hong Kong, Pokfulam
  - The Queen Mary Hospital, Hong Kong, Pokfulam

IPD SHARING:
Plan to Share IPD: No